CLINICAL TRIAL: NCT04030949
Title: Are Rectal and Genital Chlamydia Trachomatis Infections in Women Related to Anal Sex, Autoinoculation / Contamination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Napoleon Kentarchos, Residence in Dermatology and Venereology the Department of Dermatology and Venereology in Region Östergötland, Region Östergötland
Other Study IDs: 232100-0040
Record Dates: First submitted 2019-06-26; First posted 2019-07-24 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Chlamydia Trachomatis Genital Infection; Chlamydia Trachomatis Infection of Anus and Rectum
Keywords: pediatric proctoscope; oral sex,; anal sex,; MLST,; vPCR; discordance; concordance
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Secretion and epithelial cells from vaginal and rectal mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ateendes STD clinics Östergötland physician appointment: Attendees with an appointment to a physician (if she has symptoms or if she wishes a gynecological exam).
  The exam starts with an Abbot multi-collect swab taken from the anal verge, at the opening of the anal canal.
  A pediatric proctoscope (a proctoscope designed and manufactured to examine children) is used for sampling the rectal specimens using an Abbot multi-collect swab and a standard Sigma swab of Sigma virocult, followed by vaginal speculum exam. Firstly samples from the lateral fornix for wet smear are collected, secondly a swab for methylene-blue staining from the endocervical orifice followed by two Abbot multi-collect swabs for chlamydia/gonorrhoea and M.genitalium respectively from the orifice, the portio and the vaginal wall and one standard Sigma swab of Sigma virocult from the same areas. Lastly a sample is collected from the distal urethra and stained with methylene blue.
  Interventions: Other: No new interventions will be applied. MLST and MLVA even vPCR are tests already existing, tested and without any known adverse effects for the participants
- Ateendes STD clinics Östergötland, nurse appointment: The participant collects the rectal sample for chlamydia and gonorrhea (Abbot multi-collect swab) first and is instructed to try not to touch the perianal/perineal areas. Then the vaginal samples for chlamydia/gonorrhoea and M.genitalium are collected.
  There is a group of women who have been tested positive for chlamydia by self-collected vaginal swab which is sent to the patient by mail. Those are requested to attend the STD-clinic for partner tracing and are offered antibiotic treatment with doxycycline. Those accepting to participate in the study will answer the study questions and will be tested again and a nurse will collect firstly an Abbot multi-collect swab from the anal verge, at the opening of the anal canal and then two rectal swabs using a pediatric proctoscope (one Abbot multi-collect and one standard Sigma swab of Sigma virocult) and the participant will self-collect a new vaginal sample for chlamydia/gonorrhea and one for M.genitalium (two Abbot multi-collect swabs)
  Interventions: Other: No new interventions will be applied. MLST and MLVA even vPCR are tests already existing, tested and without any known adverse effects for the participants
- Ateendes STD clinics Östergötland+Jönköping partner chlamydia: Women attending the STD clinics because of a verified chlamydia infection of their current partner. This group of patients is examined and tested by a nurse or doctor before doxycycline treatment is offered.
  Those accepting to participate in the study answer the questions about the experience of receptive anal sex and fellatio (and condom use) during the last 12 months and even additional questions regarding fellatio and whether it happened that a male partner ejaculated in oral cavity of the participant.
  The first sample is an Abbot multi-collect swab taken from the anal verge and the anal canal and two more swabs are taken under the use of a pediatric proctoscope: one Abbot multi-collect and one standard Sigma swab of Sigma virocult and finally vaginal samples are collected (one Abbot multi-collect and one standard Sigma swab of Sigma virocult)
  Interventions: Other: No new interventions will be applied. MLST and MLVA even vPCR are tests already existing, tested and without any known adverse effects for the participants

INTERVENTIONS:
Other: No new interventions will be applied. MLST and MLVA even vPCR are tests already existing, tested and without any known adverse effects for the participants — No new interventions will be applied. MLST and MLVA even vPCR are tests already existing, tested and without any known adverse effects for the participants

SUMMARY:
Chlamydia trachomatis is the most common cause of sexually transmitted bacterial infection in Sweden, an infection that is notifiable according to the Communicable Diseases Act and the Communicable Diseases Ordinance.

Women account for 57 % of all cases detected since 1993. Recently published studies describe a high proportion of positive rectal chlamydia tests in women and in half of the cases there is no history of anal sex. In almost 20 % of cases, chlamydia has only been found rectally. Samples in these studies were self-collected and although the sensitivity of modern NAATs (Nucleic Acid Amplification Tests) is very high, there is even high risk of contamination of the sample due to the short anatomical distance between the vagina and the anus. Furthermore the vaginal sample has been taken prior to the rectal sample in the largest study from the Netherlands, something that further increases the risk of contamination of the rectal sample.

There are experimental animal models which support the theory that chlamydia can be transferred along the gastrointestinal tract! This is a possible explanation for the occurrence of rectal chlamydia in women who have not had anal intercourse, but it is necessary to minimize the risk of contamination.

The study will take part in three STD-clinics (2 counties) where two clinics are in the county of Östergötland (Norrköping and Linköping with totally 300 000 inhabitants) and one in the county of Jönköping (120 000 inhabitants).

The risk of contamination of the rectal samples is minimized as the rectal sample is taken first and with the use of a pediatric proctoscope (a proctoscope that is designed to examine children) which is first inserted in the anus to allow sample collection from the rectal mucosa above the pectinate line, while avoiding contact of the collecting swab with the perineal skin. Then vaginal speculum examination is performed and samples are taken from endocervix and vagina for C.trachomatis N.gonorrhoeae and M.genitalium tests. Extra samples from the anus and the vagina will be collected and immediately frozen to minus 80 degrees to allow further testing with vPCR (viability Polymerase Chain Reaction). Positive chlamydia samples will be further analyzed with a high resolution method (Multi Locus Sequence Typing, or MLST and if necessary Multi-Locus Variable number tandem repeat Analysis or MLVA) to make the discrimination of various chlamydia types possible.

DETAILED DESCRIPTION:
In the county of Östergötland.

Both STD (Sexually Transmitted Diseases) outpatient clinics in Östergötland belong to the Department of Dermatology and Venereology in Region Östergötland. The attendee has two options: either makes an appointment to a physician if the attendee has symptoms or wishes a gynecological exam because of other reasons, or make an appointment to a nurse for self-collecting tests.

All attendees answer a questionnaire including experience of receptive anal sex and fellatio (and condom use) during the last 12 months. In the study questionnaire there is an additional question regarding fellatio and whether it happened that a male partner ejaculated in her oral cavity.

At the visit by the physician:

The exam starts with an Abbot multi-collect swab taken from the anal verge, at the opening of the anal canal, where the inverstigators think the most self-taken samples come from. This sample will be immediately frozen for later analysis.

A pediatric proctoscope (a proctoscope designed and manufactured to examine children) is used for sampling the rectal specimens using an Abbot multi-collect swab and a standard Sigma swab of Sigma virocult, followed by vaginal speculum examination. Firstly samples from the lateral fornix for wet smear are collected, secondly a swab for methylene-blue staining from the endocervical orifice followed by two Abbot multi-collect swabs for chlamydia/gonorrhoea and M.genitalium respectively from the orifice, the portio and the vaginal wall and one standard Sigma swab of Sigma virocult from the same areas. Lastly a sample is collected from the distal urethra and stained with methylene blue.

Samples collected with standard Sigma swab of Sigma virocult will be immediately frozen in minus 80 grades.

Microscopic examination using a modern Zeiss microscope (Axio Lab A1) is performed. All the tubes for the chlamydia samples and the virocult samples have an extra label for the study.

All women tested with a pediatric proctoscope will answer a questionnaire about their opinion regarding this examination procedure.

At the visit by the nurse:

The participant collects the rectal sample for chlamydia/gonorrhea with an Abbot multi-collect swab first and is instructed to try not to touch the perianal/perineal areas with the swab. Then the vaginal samples for chlamydia/gonorrhoea and Mycoplasma genitalium are collected by the patient using the same type of swab.

Attendees initially not treated but turned out to have chlamydia will be asked to be tested once more to take new samples with the pediatric proctoscope before treatment is given.

Some women attend because of a verified chlamydia infection of their current partner and those are offered treatment with doxycycline. In these cases the nurse will collect first an Abbot multi-collect swab taken from the anal verge, at the opening of the anal Canal and then the rectal samples (one Abbot multi-collect swab and one standard Sigma swab of Sigma virocult) by using the pediatric proctoscope prior to the vaginal swabs which will be self-collected (one Abbot multi-collect and one standard Sigma swab of Sigma virocult).

There is another group of women who have been tested positive for chlamydia by self-collected vaginal swab which is sent to the patient by mail. Those are requested to attend the STD-clinic for partner tracing and are offered antibiotic treatment with doxycycline as standard treatment. Those accepting to participate in the study will be tested again and a nurse will collect first an Abbot multi-collect swab taken from the anal verge, at the opening of the anal canal that will be immediately frozen for later analysis and then the rectal swabs by using a pediatric proctoscope (one Abbot multi-collect and one standard Sigma swab of Sigma virocult) and the participant will collect a new vaginal sample for chlamydia/gonorrhea and one for M.genitalium (two Abbot multi-collect swabs) The first sample from the anal verge and all samples collected with standard Sigma swab of Sigma virocult will immediately be frozen to minus 80 grades for later analysis.

All samples have an extra label for the study. All women tested with a pediatric proctoscope will answer a questionnaire about their opinion regarding this examination procedure.

In the county of Jönköping:

The STD clinic of the County of Jönköping has another policy to trace and treat chlamydia trachomatis infections and the group of patients that is suitable for the study is women attending the STD clinic because of a verified chlamydia infection of their current partner. This group of patients is examined and tested by a nurse or doctor before doxycycline treatment is offered.

Those accepting to participate in the study answer the questions about the experience of receptive anal sex and fellatio (and condom use) during the last 12 months and even an additional question regarding fellatio and whether it happened that a male partner ejaculated in her oral cavity.

The exam starts with an Abbot multi-collect swab taken from the anal verge, at the opening of the anal canal. This sample will be immediately frozen for later analysis.Then the participant is tested with a pediatric proctoscope and two rectal samples are collected (one Abbot multi-collect and one standard Sigma swab of Sigma virocult) and even vaginal samples are collected at the same time (one Abbot multi-collect and one standard Sigma swab of Sigma virocult) The Abbot multi-collect swabs will be sent to Linköping for analysis. The first sample collected with Abbot multi-collect swab from the anal verge and all samples collected with standard Sigma swab of Sigma virocult will immediately be frozen to minus 80 grades for later analysis.

All samples have an extra label for the study. All women tested with a pediatric proctoscope will answer a questionnaire about their opinion regarding this procedure.

Positive chlamydia samples will be further analyzed with a high resolution method (Multi Locus Sequence Typing, or MLST and if necessary Multi-Locus Variable number tandem repeat Analysis or MLVA) to make the discrimination of various chlamydia types possible.

Discordance between chlamydial types in vagina and anus will favor the hypothesis of a currently unknown chlamydia reservoir in the anal region or a possible orogastrointestinal way of infection due to unprotected oral sex. Concordance will favor the autoinoculation of chlamydia from vagina to anus or vice versa. Moreover vPCR testing of the frozen samples will allow discrimination of real chlamydial infections (presence of viable bacteria) from contamination (presence of chlamydial DNA but not of viable bacteria). The history of oral sex and the difference in the groups that during sexual intercourse have had and have not had semen in the oral cavity may or may not strengthen the hypothesis of orogastrointestinal transport of chlamydia. After the sample collection with the pediatric proctoscope a questionnaire will be given to the attendees to investigate if the participants feel that this is an acceptable way to obtain rectal samples.

ELIGIBILITY:
Inclusion Criteria:

* All attendees at the STD clinic in the county of Östergötland
* Attendees with a verified chlamydia infection of their current partner in the county of Jönköping.

Exclusion Criteria:

* Younger than 18 years old.
* Severe rectal disease, for example, active inflammatory bowel disease or rectal cancer.
* Incapability to fill the questionnaire and / or understand the meaning / character of the study (eg women with language difficulties in Swedish, or mental development disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women above 18 years
Study Population: In the county of Östergötland all attendees at the STD clinic (the cities of Norrköping and Linköping) are offered participation consecutively.
  In the county of Jönköping women attending due to a verified chlamydia infection of their current partner.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Detection of chlamydial DNA in rectal and vaginal specimens in women attending the out-patient clinics of the county of Östergötland. | 2 years
  Detection of chlamydial DNA (NAAT) and verification of presence of viable bacteria (vPCR).Which percentage of all anogenital infections is rectal and only rectal?
Molecular typing of chlamydial DNA extracted from specimens from vaginal and rectal mucosa. Frequency of concordance or discordance between chlamydial types found in respective site. | 2 years
  Molecular typing (MLST and if needed MLVA) of chlamydial DNA in participants with simultaneous infection of the vagina and the rectum. Number of participants with simultaneous vaginal and rectal chlamydial infections with the same chlamydial type in both sites (concordance) vs number of participants with simultaneous vaginal and rectal chlamydial infections with different chlamydial type in vagina and rectum (discordance).
Incidence of true rectal chlamydial infections in women not practicing anal sex. Is there statistically significant difference between those that practice fellatio or not and those that have received sperma orally or not? | 2 years
  Among participants with positive rectal chlamydial tests there will exist a subgroup not practicing anal sex according to the results of previous studies. If the theory of orogastrointestinal proliferation is possible in humans, then among those women there should be a number practicing fellatio and the number of those receiving sperm orally could more often have a rectal infection.
Chlamydia infection specificity of swabs taken without proctoscope vs swabs taken with pediatric proctoscope. Risk for false positive for swabs taken with and without pediatric proctoscope. | 2 years
  How many positive rectal chlamydia tests are verified as true infections with a positive vPCR and how many positive rectal chlamydia tests are a result of DNA contamination? Which is the true sensitivity of self-taken rectal tests and how often are self-taken tests false positive?
Grade of discomfort and willingness of participants to undergo rectal sampling with a pediatric proctoscope. | 2 years
  All participants will be asked to fill a standard questionnaire after the proctoscopy. The grade of discomfort will be assessed by each participant with the help of a Visual Analogue Scale (VAS), where the one end is equal to no discomfort and the other is equal to the worst discomfort experienced.
  The willingness of the participants to take the rectal tests the same way in the future if requested will be assessed by each participant again with the help of a Visual Analogue Scale, where then one end is equal to willing to take the rectal tests the same way again, while the other end equal to not willing.
  Both scales will consist of 100 mm long lines and the results will be measured according to the intervals of 0-4 mm (no discomfort/willing), 5-44 mm (mild discomfort/probably willing), 45-74 mm (moderate discomfort/probably not willing) and 75-100 mm (severe discomfort/ not willing).

SECONDARY OUTCOMES:
Frequency of symptoms in patients with a rectal chlamydial infection. | 2 years
  Frequency of symptoms in patients with a rectal chlamydial infection. How often do participants with rectal chlamydia infection experience symptoms?
Comparison of chlamydial bacterial loads measured in chlamydia copies per milliliter between rectal and vaginal specimens. | 2 years
  Using quantitative PCR we will compare the chlamydial bacterial load between vaginal and rectal infections, measured as chlamydia copies per milliliter given a less effective inflammatory reaction in the rectal mucosa
Prevalence of non-specific cervicitis among participants with rectal chlamydial infections vs participants without rectal chlamydial infections. | 2 years
  A possible explanation for non-specific vaginitis is a rectal chlamydial infection/reservoir that can proliferate to the vagina via autoinoculation.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Falk, Assistant Professor, Study Director — Region Östergötland
Locations (2):
- Sweden (2):
  - Department of Dermatology and Venereology in Region Östergötland, Linköping, County of Östergötland
  - Department of Dermatology and Venereology in the county of Jönköping, Jönköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Falk L. The overall agreement of proposed definitions of mucopurulent cervicitis in women at high risk of Chlamydia infection. Acta Derm Venereol. 2010 Sep;90(5):506-11. doi: 10.2340/00015555-0924. PMID 20814628
- [Result] Taylor SN. Cervicitis of unknown etiology. Curr Infect Dis Rep. 2014 Jul;16(7):409. doi: 10.1007/s11908-014-0409-x. PMID 24859465
- [Result] Klint M, Fuxelius HH, Goldkuhl RR, Skarin H, Rutemark C, Andersson SG, Persson K, Herrmann B. High-resolution genotyping of Chlamydia trachomatis strains by multilocus sequence analysis. J Clin Microbiol. 2007 May;45(5):1410-4. doi: 10.1128/JCM.02301-06. Epub 2007 Feb 28. PMID 17329456
- [Result] Andersson N, Boman J, Nylander E. Rectal chlamydia - should screening be recommended in women? Int J STD AIDS. 2017 Apr;28(5):476-479. doi: 10.1177/0956462416653510. Epub 2016 Jul 10. PMID 27235696
- [Result] van Liere GAFS, Dukers-Muijrers NHTM, Levels L, Hoebe CJPA. High Proportion of Anorectal Chlamydia trachomatis and Neisseria gonorrhoeae After Routine Universal Urogenital and Anorectal Screening in Women Visiting the Sexually Transmitted Infection Clinic. Clin Infect Dis. 2017 Jun 15;64(12):1705-1710. doi: 10.1093/cid/cix243. PMID 28369227
- [Result] Schachter J, Grossman M, Sweet RL, Holt J, Jordan C, Bishop E. Prospective study of perinatal transmission of Chlamydia trachomatis. JAMA. 1986 Jun 27;255(24):3374-7. PMID 3712696
- [Result] Rank RG, Yeruva L. Hidden in plain sight: chlamydial gastrointestinal infection and its relevance to persistence in human genital infection. Infect Immun. 2014 Apr;82(4):1362-71. doi: 10.1128/IAI.01244-13. Epub 2014 Jan 13. PMID 24421044
- [Result] Carre H, Edman AC, Boman J, Nylander E. Chlamydia trachomatis in the throat: is testing necessary? Acta Derm Venereol. 2008;88(2):187-8. doi: 10.2340/00015555-0382. No abstract available. PMID 18311460
- [Result] Sethupathi M, Blackwell A, Davies H. Rectal Chlamydia trachomatis infection in women. Is it overlooked? Int J STD AIDS. 2010 Feb;21(2):93-5. doi: 10.1258/ijsa.2008.008406. Epub 2009 Nov 16. PMID 19917639
- [Result] Foschi C, Salvo M, Cevenini R, Marangoni A. Chlamydia trachomatis antimicrobial susceptibility in colorectal and endocervical cells. J Antimicrob Chemother. 2018 Feb 1;73(2):409-413. doi: 10.1093/jac/dkx392. PMID 29077843
- [Result] Herrmann B, Isaksson J, Ryberg M, Tangrot J, Saleh I, Versteeg B, Gravningen K, Bruisten S. Global Multilocus Sequence Type Analysis of Chlamydia trachomatis Strains from 16 Countries. J Clin Microbiol. 2015 Jul;53(7):2172-9. doi: 10.1128/JCM.00249-15. Epub 2015 Apr 29. PMID 25926497
- See also: Related Info — http://mlstdb.bmc.uu.se/